CLINICAL TRIAL: NCT03899935
Title: Feasibility and Safety of Endometriosis Laparoscopic Removal in Obese Patients: a Propensity Score Method Analysis
Brief Title: Laparoscopy for Endometriosis in Obese Patients
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Renato Seracchioli, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: ObesityEndometriosis
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Endometriosis; Obesity
Keywords: Endometriosis; Obesity; Laparoscopy
MeSH Terms: conditions — Endometriosis; Obesity | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: obese patients: Obese patients undergoing laparoscopic surgery for endometriosis
  Interventions: Procedure: Laparoscopy
- Group B: non-obese patients: Non-obese patients undergoing laparoscopy for endometriosis
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Laparoscopy for endometriosis

SUMMARY:
Evaluation of surgical outcomes of endometriosis laparoscopic surgery in obese patients.

DETAILED DESCRIPTION:
Obesity may influence surgical variables such as operative time, laparotomic conversion rate and intraoperative and postoperative complication rate. Moreover, it might influence the hospital length of stay. For that reason, the study aims to compare a group of obese patients with a non-obese group of patients about these topics.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients undergoing endometriosis laparoscopic treatment
* Obteined Informed Consensus

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive patients affected by endometriosis undergoing to laparoscopic endometriosis removal.
Sampling Method: Probability Sample
Enrollment: 1230 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Operative time | Intraoperative: from the skin incision to the skin suture
  Comparison of operative time, expressed in minutes, between Group A and Group B

SECONDARY OUTCOMES:
Laparotomic conversion rate | Intraoperative
  Comparison of laparotomic conversion rate between Group A and Group B
Hospital length of stay | Postoperative: from surgery to hospitalization discharge, assessed up to 30 days after surgery.
  Comparison of hospital length of stay, expressed in days, between Group A and Group B
Intraoperative complication rate | Intraoperative
  Comparison of intraoperative complication rate between Group A and Group B. Intraoperative complication rate is assessed using Clavien-Dindo Classification (from grade I to V, where I means any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions, and V means the death of a patient)
Postoperative complication rate | Postoperative: from surgery to hospitalization discharge, assessed up to 30 days after surgery.
  Comparison of postoperative complication rate between Group A and Group B. Postoperative complication rate is assessed using Clavien-Dindo Classification (from grade I to V, where I means any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions, and V means the death of a patient)

CONTACTS AND LOCATIONS:
Locations (1):
- Diego Raimondo, Bologna, BO, Italy